CLINICAL TRIAL: NCT00921700
Title: Analgesic Effect of Ibuprofen 400 mg/Paracetamol 1000 mg, Ibuprofen 400 mg/ Paracetamol 1000 mg/60 mg Codeine, and Paracetamol 1000 mg/Codeine 60 mg: A Single-dose, Randomized, Placebo-controlled and Double-blind Study
Brief Title: Analgesic Effect of Paracetamol, Paracetamol + Codeine, Ibuprofen and Their Combination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Lasse Ansgar Skoglund, Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PARIBU-022; EUDRACT No. 2007-001778-10
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Pain, Postoperative
Keywords: Paracetamol; Acetaminophen; Ibuprofen; Pain; Postoperative pain; third molar
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ibuprofen; Acetaminophen; Codeine; acetaminophen, codeine drug combination; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ibuprofen + Paracetamol (Experimental): Single oral dose of ibuprofen 400 mg + paracetamol (acetaminophen) 1000 mg
  Interventions: Drug: Ibuprofen + Paracetamol
- Ibuprofen + Paracetamol + Codeine (Experimental): Single oral dose of ibuprofen 400 mg + paracetamol (acetaminophen) 1000 mg + codeine 60 mg
  Interventions: Drug: Ibuprofen + Paracetamol + Codeine
- Paracetamol + Codeine (Active Comparator): Single oral dose of paracetamol (acetaminophen) 1000 mg + codeine 60 mg
  Interventions: Drug: Paracetamol + Codeine
- Placebo (Placebo Comparator): Single oral dose of lactose as placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen + Paracetamol — Single oral dose of ibuprofen 400 mg combined with paracetamol (acetaminophen) 1000 mg in gelatine capsules
  Other Names: Ibuprofen; ATC code: M01A E01; Paracetamol (Acetaminophen); ATC code: N02B E01
  Arms: Ibuprofen + Paracetamol
Drug: Ibuprofen + Paracetamol + Codeine — Single oral dose of ibuprofen 400 mg combined with paracetamol (acetaminophen) 1000 mg and codeine 60 mg in gelatine capsules
  Other Names: Ibuprofen; ATC code: M01A E01; Paracetamol (Acetaminophen); ATC code: N02B E01; Codeine; ATC code: R05D A04
  Arms: Ibuprofen + Paracetamol + Codeine
Drug: Paracetamol + Codeine — Single oral dose of paracetamol (acetaminophen) 1000 mg combined with codeine 60 mg in gelatine capsules
  Other Names: Paracetamol (Acetaminophen); ATC code: N02B E01; Codeine; ATC code: R05D A04
  Arms: Paracetamol + Codeine
Drug: Placebo — Single oral dose of lactose as placebo in gelatine capsules
  Other Names: Lactose; CAS No: 63-42-3
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the combination of paracetamol (acetaminophen) and other NSAIDs with or without weak opioids can give synergistic analgesic effect.

DETAILED DESCRIPTION:
Combining paracetamol and other NSAIDs could give a theoretical synergistic analgesic effect according to already known or assumed mechanisms of action. Synergism is defined as an additive or supra-additive effect not achieved by one of the drugs alone. Such synergism is shown in clinical studies between acetaminophen and naproxen in coxarthrosis and rheumatoid arthritis. Later, a significant additive effect of 100 mg diclofenac with 1 g acetaminophen was demonstrated in a dental pain model.

One review article conclude that acetaminophen and NSAIDs may be appropriate to combine, and the combination is superior to acetaminophen, but not to NSAIDs alone. This view is contested by another review article which concludes that paracetamol may enhance the analgesic effect when added to an NSAID. In both reviews the authors also state that the clinical trials are too few, with different drug formulations, and different pain models not allowing definite conclusions.

There seems to be a need for studies investigating the potential synergistic effects of paracetamol combined with another NSAID displaying similar pharmacokinetic characteristics. To the best of our knowledge no published study has investigated the analgesic effect of the combination of ibuprofen and paracetamol, ibuprofen and paracetamol + codeine versus placebo (i.e. negative control to adjust for possible analgesic placebo effects) and the best standard analgesic treatment (i.e. paracetamol + codeine) as a positive control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients of ASA class I in need of surgical removal of impacted third molars and with at least moderate postoperative pain as defined by subjective score on a verbal rating scale after surgical removal of third molars.

Exclusion Criteria:

* Females stating not suspected or not verified pregnancy after being questioned by investigator.
* Patients who have used analgesics for 3 days prior to the day of surgery.
* Patients with known active gastrointestinal bleeding or ulcer.
* Patients with any known hypersensitivity to NSAIDs.
* Patients with other drug treatment than contraceptives.
* Patients smoking before taking the test-drug or during the observation period.
* Drug addicts or rehabilitated drug addicts.
* Patients with surgery time exceeding 60 minutes
* Peroperative complications such as profuse bleeding or perforation to the maxillary sinus requiring additional drug treatment during or after the surgical removal of the third molar.
* Postoperative complications such as extended bleeding, nausea and regurgitation during the observation period.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2009-06; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Sum pain intensity SPI (0-10 Numerical Rating Scale) | 6 hours

SECONDARY OUTCOMES:
Sum pain intensity difference score (PID) | 6 hours
Overall assessment of efficacy (4-point Verbal Rating Scale) | 6 hours
Adverse effects AE (Specific reporting of AE - type, duration and severity) | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lasse A Skoglund, DDS, DSci, Study Director — University of Oslo; Gaute Lyngstad, DDS, Principal Investigator — University of Oslo
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Background] Seideman P. Additive effect of combined naproxen and paracetamol in rheumatoid arthritis. Br J Rheumatol. 1993 Dec;32(12):1077-82. doi: 10.1093/rheumatology/32.12.1077. PMID 8252318
- [Background] Seideman P, Samuelson P, Neander G. Naproxen and paracetamol compared with naproxen only in coxarthrosis. Increased effect of the combination in 18 patients. Acta Orthop Scand. 1993 Jun;64(3):285-8. doi: 10.3109/17453679308993626. PMID 8322582
- [Background] Breivik EK, Barkvoll P, Skovlund E. Combining diclofenac with acetaminophen or acetaminophen-codeine after oral surgery: a randomized, double-blind single-dose study. Clin Pharmacol Ther. 1999 Dec;66(6):625-35. doi: 10.1053/cp.1999.v66.103629001. PMID 10613619
- [Background] Romsing J, Moiniche S, Dahl JB. Rectal and parenteral paracetamol, and paracetamol in combination with NSAIDs, for postoperative analgesia. Br J Anaesth. 2002 Feb;88(2):215-26. doi: 10.1093/bja/88.2.215. PMID 11878655
- [Background] Hyllested M, Jones S, Pedersen JL, Kehlet H. Comparative effect of paracetamol, NSAIDs or their combination in postoperative pain management: a qualitative review. Br J Anaesth. 2002 Feb;88(2):199-214. doi: 10.1093/bja/88.2.199. PMID 11878654
- [Background] Skoglund LA, Skjelbred P, Fyllingen G. Analgesic efficacy of acetaminophen 1000 mg, acetaminophen 2000 mg, and the combination of acetaminophen 1000 mg and codeine phosphate 60 mg versus placebo in acute postoperative pain. Pharmacotherapy. 1991;11(5):364-9. PMID 1745622
- [Derived] Lyngstad G, Skjelbred P, Swanson DM, Skoglund LA. Analgesic effect of oral paracetamol 1000 mg/ibuprofen 400 mg, paracetamol 1000 mg/codeine 60 mg, paracetamol 1000 mg/ibuprofen 400 mg/codeine 60 mg, or placebo on acute postoperative pain: a single-dose, randomized, and double-blind study. Eur J Clin Pharmacol. 2023 Aug;79(8):1131-1141. doi: 10.1007/s00228-023-03525-0. Epub 2023 Jun 22. PMID 37349498